CLINICAL TRIAL: NCT01121094
Title: Fetal Parenchymatic Evaluation (Liver, Spleen) Using T2* Sequences.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sheba Medical Center, Sheba Medical Center
Other Study IDs: SHEBA-09-7502-OG-SMC
Record Dates: First submitted 2010-05-09; First posted 2010-05-12 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Iron Overload
Keywords: Liver, spleen , T2* , MRI, fetus
MeSH Terms: conditions — Iron Overload

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to prospectively evaluated the T2* values of normal feti.A standardized scale of T2* values for fetal and neonatal iron organ overload have yet to be reported or devised.

DETAILED DESCRIPTION:
The purpose of this study is to prospectively evaluate the T2* values of normal feti. This study will be offered to mothers undergoing fetal MRI for any indication. Subjects will be required to sign an informed consent from. The addition of T2* sequences will add 2-4 minutes to the whole scan, not exposing the mother or the fetus to ionizing radiation or the administration of contrast material. A standardized scale has been created and multi-center studies have been conducted using different vendor scanners in order to verify the consistency of these scale. T2 and T2* sequences have been addressed anecdotally in the literature as non invasive options for the evaluation fetal iron deposition . However, a standardized scale of T2* values for fetal and neonatal iron organ overload have yet to be reported or devised.

ELIGIBILITY:
Inclusion Criteria:

* Any MRI study for fetus

Exclusion Criteria:

* Known iron deposition problem in the mother of fetus

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will be offered to motheres undergoing fetal MRI for any indication.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba medical center, Tel Litwinsky, Israel, Israel